CLINICAL TRIAL: NCT06497660
Title: Effect of Neoadjuvant Chemotherapy on Cardiac Function of Perioperative Patients With Breast Cancer and New Strategies for Anesthesia Response: a Multicenter, Prospective, Randomized, Controlled Study
Brief Title: Effect of Neoadjuvant Chemotherapy on Cardiac Function of Perioperative Patients With Breast Cancer and New Strategies for Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LZMLRJXFZHLRXAYJ
Record Dates: First submitted 2024-05-05; First posted 2024-07-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy; Perioperative Period; Anaesthesia; Cardiac Function
MeSH Terms: conditions — Breast Neoplasms | interventions — Deoxyepinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- A α group (Experimental): Breast cancer patients with neoadjuvant chemotherapy scheme of "EC-T" and selective surgery were selected, and they were intervened with norepinephrine during the perioperative period.
  Interventions: Drug: Deoxyadrenaline
- B α group (Experimental): Breast cancer patients with "TCb" neoadjuvant chemotherapy and elective surgery were selected, and they were intervened with norepinephrine during the perioperative period
  Interventions: Drug: Deoxyadrenaline
- C α group (Experimental): Breast cancer patients with "TCbHP" neoadjuvant chemotherapy and elective surgery were selected, and they were intervened with norepinephrine during the perioperative period.
  Interventions: Drug: Deoxyadrenaline
- control α group (Placebo Comparator): Patients with breast cancer who have not received neoadjuvant chemotherapy and who have undergone elective surgery, and who have received perioperative intervention with norepinephrine.
  Interventions: Drug: Deoxyadrenaline
- A β group (Experimental): Select breast cancer patients with neoadjuvant chemotherapy scheme of "EC-T" and elective surgery, and use normal saline for control during perioperative period.
  Interventions: Drug: normal saline
- B β group (Experimental): Breast cancer patients with "TCb" neoadjuvant chemotherapy and elective surgery were selected, and physiological saline was used as control during perioperative period.
  Interventions: Drug: normal saline
- C β group (Experimental): Breast cancer patients with "TCbHP" neoadjuvant chemotherapy and elective surgery were selected, and physiological saline was used as control during perioperative period.
  Interventions: Drug: normal saline
- control β group (Placebo Comparator): Breast cancer patients who have not received neoadjuvant chemotherapy and who have undergone elective surgery, and who use normal saline control during the perioperative period.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Deoxyadrenaline — Deoxyadrenaline is a vasoactive drug
  Arms: A α group; B α group; C α group; control α group
Drug: normal saline — Deoxyadrenaline is a vasoactive drug
  Arms: A β group; B β group; C β group; control β group

SUMMARY:
As is well known, perioperative hemodynamic fluctuations, such as decreased blood pressure and heart rate, and cardiac dysfunction, are common complications after anesthesia. General anesthetics such as propofol and sufentanil can inhibit the central nervous system, reduce cardiac excitability and myocardial contractility, dilate peripheral blood vessels, and have a high incidence of hypotension, especially during anesthesia induction, which is particularly common in the elderly and those with underlying underlying diseases before surgery.

However, the current research on the impact of neoadjuvant chemotherapy on perioperative cardiac function in patients is not specific, and there is no unified anesthesia strategy for these effects during the perioperative period. Therefore, this study aims to explore: 1. the effect of neoadjuvant chemotherapy on perioperative cardiac function in patients; 2. Improve the anesthesia plan and further explore new strategies for perioperative organ protection for such patients. The research design is a prospective, randomized, controlled trial.

DETAILED DESCRIPTION:
Traditional chemotherapy is a common treatment for cancer, usually performed after surgery, with the aim of assisting in the removal of remaining cancer cells. Nausea, vomiting, fatigue, hair loss, bone marrow suppression, and other common complications can even affect the function of important organs such as the heart, lungs, and brain. In the 1980s, with the reflection on traditional chemotherapy and further understanding of tumor biology, clinical trials and research began to focus on a method of neoadjuvant chemotherapy that combines surgical resection before surgery.

Neoadjuvant chemotherapy refers to the systemic chemotherapy performed before implementing local treatment methods (such as surgery), with the aim of reducing the size of the tumor, killing invisible metastatic cells early, and reducing adverse reactions to traditional chemotherapy [6], which is a new chemotherapy method that is beneficial for subsequent surgery, radiotherapy, and other treatments. However, it should be noted that neoadjuvant chemotherapy may still cause a certain degree of cardiac dysfunction.

As is well known, perioperative hemodynamic fluctuations, such as decreased blood pressure and heart rate, and cardiac dysfunction, are common complications after anesthesia. General anesthetics such as propofol and sufentanil can inhibit the central nervous system, reduce cardiac excitability and myocardial contractility, dilate peripheral blood vessels, and have a high incidence of hypotension, especially during anesthesia induction, which is particularly common in the elderly and those with underlying underlying diseases before surgery.

In summary, after completing neoadjuvant chemotherapy, the patient's physical and mental functions are affected to a certain extent. If combined with the effects of anesthetic drugs, the hemodynamic fluctuations are greater than those of the general population, which may further cause cardiac dysfunction and is worthy of attention. However, the current research on the impact of neoadjuvant chemotherapy on perioperative cardiac function in patients is not specific, and there is no unified anesthesia strategy for these effects during the perioperative period. Therefore, this study aims to explore: 1. the effect of neoadjuvant chemotherapy on perioperative cardiac function in patients; 2. Improve the anesthesia plan and further explore new strategies for perioperative organ protection for such patients. The research design is a prospective, randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above;
2. Left ventricular ejection fraction shall not be less than 45% before neoadjuvant chemotherapy and not less than 40% after neoadjuvant chemotherapy;
3. The electrocardiogram shows sinus rhythm;
4. Acetylsalicylic acidlevel I to III;
5. Can understand and cooperate with the research process.

Exclusion Criteria:

1. Patients with congenital organic heart disease, arrhythmia requiring intervention, heart valve disease, cardiomyopathy, high atrioventricular and bundle branch block, history of myocardial infarction, severe hypertension, long-term diabetes and other diseases affecting heart function;
2. Patients with severe dysfunction of important organs such as liver and kidney, who are intolerant to neoadjuvant chemotherapy or surgical anesthesia;
3. Patients who are allergic to the drugs used in this study;
4. Patients with mental illness, consciousness disorders, and communication barriers;
5. Patients with severe coagulation dysfunction;
6. Patients who have used monoamine oxidase inhibitors within two weeks prior to anesthesia surgery;
7. Patients who refused to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-02 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The degree of blood pressure decrease during anesthesia induction | On the day of surgery, compare the blood pressure changes of patients after entering the operating room and anesthesia induced tracheal intubation, with a maximum of 12 months after surgery.
  Compare the blood pressure changes of patients after entering the operating room and undergoing anesthesia induced tracheal intubation.（Unit in mmHg）

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Affiliated Union Hospital, Fuzhou, Fujian, China